CLINICAL TRIAL: NCT02565615
Title: ATORVASTATIN EFFECTIVENESS AND SAFETY IN CARDIOLOGY PATIENTS IN REAL WORLD SETTING: A REGISTRY STUDY IN CHINA
Brief Title: Atorvastatin Effectiveness and Safety in Cardiology Patients in Real World Setting
Acronym: ATTENTION
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581197
Record Dates: First submitted 2015-09-15; First posted 2015-10-01 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease, Hypercholesterolemia, Hypertension
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atorvastatin dose titration (single-arm): Judged by investigators, patients in cardiology department who are using atorvastatin can be included into this study, if they are eligible. During the study, the dose can be titrated based on the judgement of investigator
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Because this is a non-interventional study, there is no intervention here.

SUMMARY:
The study is to verify atorvastatin effectiveness and safety in Chinese population, and explore the optimal atorvastatin regimens in high-to-moderate risk for ASCVD。

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years;
* Cardiology patients who has been prescribed atorvastatin by physician's clinical judgment under normal clinical care. These patients will include those with established coronary heart disease, or having multiple risk factors and at risk for cardiovascular disease, or primary hypercholesterolemia.
* Baseline laboratory reports prior to starting atorvastatin therapy can be tracked , including lipid measurement, liver function, and Creatine Kinase (CK) value. The date of baseline reports should be within 1 month before taking atorvastatin or within 24h after starting atorvastatin therapy.
* Evidence of a personally or his/her legally acceptable representative signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study and accept follow-up visit.

Exclusion Criteria:

* Patients who have regularly taken atorvastatin therapy more than 4 weeks before enrollment
* Concomitant any other lipid-lower medication at baseline, or during the study conduction on physician clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese cardiology patients
Sampling Method: Non-Probability Sample
Enrollment: 5115 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- China (54):
  - First People's Hospital of Fuyang City, Fuyang, Anhui
  - China Meitan General Hospital, Beijing, Beijing Municipality
  - CHINA-JAPAN Friendship Hospital, Beijing, Beijing Municipality
  - Fu Xing Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - NAVY General Hospital, Beijing, Beijing Municipality
  - Guang'anmen hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District , Beijing, Beijing, Beijing Municipality
  - People's Hospital of Beijing Daxing District, Beijing, Beijing Municipality
  - China Meitan General Hospital, Biejing, Beijing Municipality
  - Chongqing Dianjiang People's Hospital, Chongqing, Chongqing Municipality
  - Yongchuan hospital of chongqing medical university, Chongqing, Chongqing Municipality
  - Chongqing Wanzhou People's Hospital, Chongqing, Chongqing Municipality
  - Fuling center hospital of chongqing city, Chongqing, Chongqing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen, Fujian
  - Shunde people's Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The Second Hospital of Hebei University, Shijiazhuang, Hebei
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The Peoples Hspital of Hebi City, Hebi, Henan
  - Jiaozuo City Second People's Hospital, Jiaozuo, Henan
  - Puyang Oilfield General Hosipital, Puyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The first affiliated hospital of henan university of TCM, Zhengzhou, Henan
  - Zhengzhou No. 7 People's Hospital, Zhengzhou, Henan
  - Wuhan University - Renmin Hospital (Hubei General Hospital), Wuhan, Hubei
  - Huai'An First People's Hospital, Huaian, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangning People's Hospital, Nanjing, Jiangsu China
  - Cardiology Provincial Hospital of Jiangsu Province, Nanjing, Jiangsu,china
  - Nanjing colleague hospital, Nanjing, Jiangsu，china
  - The 2nd hospital of Nanchang university, Nanchang, Jiangxi
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Nanjing Red Cross Hospital, Nanjing, Nanjing, Jiangsu
  - Ji'nan Central Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai University of Traditional Chinese Medicine affiliated Yueyang Hospital of traditional Chine, Shanghai, Shanghai，china
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Dongyang People's Hospital, Jinhua, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The Affiliated Hospital of Medical College of Ningbo University, Ningbo, Zhejiang
  - Quzhou Hospital of Zhejiang University, Quzhou, Zhejiang
  - Ruian People's Hospital, Ruian, Zhejiang
  - The first people's Hospital of Xiaoshan District, Hangzhou, Zhejiang China
  - Lanxi Municipal People's Hospital, Lanxi, Zhejiangchina
  - Beijing Anzhen Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Hospital attached to aeromedicine institute of P.L.A (466 Hospital), Beijing
  - Shanghai Yangpu District Central Hospital, Shanghai
  - Shanghai Minhang District Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A2581197

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin <=10 mg: Participants received Atorvastatin <=10 mg daily according to doctor's prescription.
- Atorvastatin 20 mg: Participants received Atorvastatin 20 mg daily according to doctor's prescription.
- Atorvastatin 30 mg: Participants received Atorvastatin 30 mg daily according to doctor's prescription.
- Atorvastatin 40 mg: Participants received Atorvastatin 40 mg daily according to doctor's prescription.
- Atorvastatin Unknown Dosage: Participants didn't complete dosing information including dosing page recording 'NOT DONE', or missing Week 12 dosing event, or records with missing stop date of dosing.
Period: Overall Study
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Started | 291 | 3080 | 21 | 101 | 1622
Treated | 291 | 3080 | 21 | 101 | 1055
Completed | 288 | 3044 | 21 | 98 | 21
Not Completed | 3 | 36 | 0 | 3 | 1601
Not completed — Death | 0 | 1 | 0 | 0 | 4
Not completed — Not willing to participate in study | 2 | 21 | 0 | 1 | 169
Not completed — Lost to Follow-up | 0 | 4 | 0 | 1 | 765
Not completed — Not meeting eligibility criteria | 0 | 7 | 0 | 0 | 25
Not completed — Reason not defined | 0 | 2 | 0 | 1 | 62
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 9
Not completed — Untreated | 0 | 0 | 0 | 0 | 567

BASELINE CHARACTERISTICS:
Population: Included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage | Total
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055 | 4548
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (12.0) | 61.3 (11.6) | 59.5 (8.4) | 63.2 (11.3) | 62.2 (12.3) | 61.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 1390 | 11 | 39 | 483 | 2067
  Male | 147 | 1690 | 10 | 62 | 572 | 2481
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] — Population: Included participants with non-missing values
  kg
    number analyzed (Participants) | 282 | 3029 | 21 | 98 | 1026 | 4456
    (all) | 64.9 (11.0) | 67.9 (11.8) | 68.6 (8.2) | 67.5 (11.4) | 66.0 (12.2) | 67.3 (11.9)
Height [Mean (Standard Deviation); unit: cm] — Population: Included participants with non-missing values
  cm
    number analyzed (Participants) | 282 | 3035 | 21 | 98 | 1024 | 4460
    (all) | 163.3 (7.8) | 164.6 (7.8) | 166.0 (6.9) | 163.8 (8.4) | 164.1 (7.7) | 164.4 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Achievement Rate for Low Density Lipoprotein-Cholesterol (LDL-C) for Overall
Description: Achievement Rate was defined as ratio of number of participants who achieved LDL-C target value to number of participants who completed 12-week follow up.
Time Frame: 12 weeks
Population: The full analysis set (FAS) analysis population included all enrolled in the study that received at least 1 dose of atorvastatin and completed 12- week follow-up. "Atorvastatin Unknown Dosage" arm did not meet FAS criteria.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
Ratio | 0.79 [0.716 to 0.857] | 0.67 [0.640 to 0.690] | 0.83 [0.359 to 0.996] | 0.57 [0.432 to 0.698]

2. Primary Outcome: Achievement Rate for LDL-C by Dose Group Within Each Cardiovascular Disease (CVD) Risk Level
Description: Achievement Rate was defined as ratio of number of participants who achieved LDL-C target value to number of participants who completed 12-week follow up according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: 12 weeks
Population: The full analysis set (FAS) analysis population included all enrolled in the study that received at least 1 dose of atorvastatin and completed 12- week follow-up. "Atorvastatin Unknown Dosage" arm did not meet FAS criteria. Number analyzed refers to number of participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
Ratio
  Low risk: number analyzed (Participants) | 13 | 129 | 0 | 2
  Low risk | 1.00 [0.735 to 1.000] | 0.93 [0.870 to 0.967] |  | 1.00 [0.158 to 1.000]
  Moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Moderate risk | 1.00 [0.839 to 1.000] | 0.89 [0.827 to 0.936] |  | 0.78 [0.400 to 0.972]
  High risk: number analyzed (Participants) | 88 | 733 | 6 | 25
  High risk | 0.77 [0.671 to 0.855] | 0.68 [0.649 to 0.718] | 0.83 [0.359 to 0.996] | 0.56 [0.349 to 0.756]
  Very High risk: number analyzed (Participants) | 19 | 438 | 0 | 22
  Very High risk | 0.53 [0.289 to 0.756] | 0.48 [0.432 to 0.529] |  | 0.45 [0.244 to 0.678]

3. Secondary Outcome: Change From Baseline for Lipid Parameters at Week 12 for Overall
Description: Lipid parameters included LDL-C, High-Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol (TC), and Triglycerides (TG). The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from Baseline data was reported.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
milligram/deciliter (mg/dL)
  Cholesterol: number analyzed (Participants) | 139 | 1410 | 6 | 56
  Cholesterol | -24.81 (43.971) | -45.12 (394.177) | -40.35 (44.527) | -36.98 (54.175)
  Cholesterol (HDL): number analyzed (Participants) | 139 | 1409 | 6 | 56
  Cholesterol (HDL) | 0.55 (10.619) | 0.44 (13.643) | 0.13 (7.421) | -0.17 (8.493)
  Cholesterol (LDL): number analyzed (Participants) | 139 | 1407 | 6 | 56
  Cholesterol (LDL) | -25.26 (35.375) | -31.47 (38.285) | -31.40 (34.152) | -36.00 (40.783)
  Triglycerides: number analyzed (Participants) | 139 | 1409 | 6 | 56
  Triglycerides | -2.69 (94.228) | -27.55 (107.785) | -83.19 (151.512) | -20.97 (160.296)

4. Secondary Outcome: Percent Change From Baseline for Lipid Parameters at Week 12 for Overall
Description: Lipid parameters included LDL-C, High-Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol (TC), and Triglycerides (TG). The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Percent change from baseline was reported.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change (%)
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
Percent Change (%)
  Cholesterol: number analyzed (Participants) | 139 | 1410 | 6 | 56
  Cholesterol | -9.96 (24.219) | -13.66 (34.091) | -17.33 (19.989) | -3.07 (104.388)
  Cholesterol (HDL): number analyzed (Participants) | 139 | 1409 | 6 | 56
  Cholesterol (HDL) | 3.68 (26.013) | 4.18 (25.386) | 1.52 (15.985) | 0.91 (15.835)
  Cholesterol (LDL): number analyzed (Participants) | 139 | 1407 | 6 | 56
  Cholesterol (LDL) | -17.40 (32.437) | -20.11 (50.643) | -22.57 (26.524) | -23.68 (25.476)
  Triglycerides: number analyzed (Participants) | 139 | 1409 | 6 | 56
  Triglycerides | 12.03 (82.582) | -4.04 (52.636) | -27.55 (33.921) | -12.33 (34.679)

5. Secondary Outcome: Change From Baseline for Lipid Parameters at Week 12 Within Each CVD Risk Group
Description: Lipid parameters included LDL-C, High-Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol (TC), and Triglycerides (TG) according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes. The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from baseline data was reported.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
mg/dL
  Cholesterol-Low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Cholesterol-Low risk | -51.42 (42.967) | -47.99 (56.938) |  | -94.98 (71.530)
  Cholesterol-Moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol-Moderate risk | -26.97 (42.807) | -43.23 (49.231) |  | -5.28 (61.380)
  Cholesterol- High risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Cholesterol- High risk | -27.04 (43.996) | -56.59 (552.696) | -40.35 (44.527) | -38.43 (49.029)
  Cholesterol- Very high risk: number analyzed (Participants) | 19 | 426 | 0 | 22
  Cholesterol- Very high risk | 4.63 (31.528) | -25.78 (49.060) |  | -43.16 (51.923)
  Cholesterol (HDL)- Low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Cholesterol (HDL)- Low risk | -0.29 (8.445) | -1.80 (9.943) |  | -8.30 (24.298)
  Cholesterol (HDL)- Moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol (HDL)- Moderate risk | 1.27 (10.964) | -0.92 (10.398) |  | 5.06 (10.908)
  Cholesterol (HDL)- High risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Cholesterol (HDL)- High risk | 0.18 (11.112) | 0.64 (14.169) | 0.13 (7.421) | 1.21 (5.473)
  Cholesterol (HDL)- Very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Cholesterol (HDL)- Very high risk | 1.99 (9.675) | 1.25 (14.585) |  | -3.02 (7.447)
  Cholesterol (LDL)- Low risk: number analyzed (Participants) | 12 | 127 | 0 | 2
  Cholesterol (LDL)- Low risk | -49.29 (37.689) | -42.37 (37.719) |  | -74.71 (53.238)
  Cholesterol (LDL)- Moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol (LDL)- Moderate risk | -26.07 (33.338) | -37.50 (37.162) |  | -25.91 (32.562)
  Cholesterol (LDL)- High risk: number analyzed (Participants) | 87 | 710 | 6 | 23
  Cholesterol (LDL)- High risk | -26.61 (35.093) | -33.10 (39.149) | -31.40 (34.152) | -34.61 (44.918)
  Cholesterol (LDL)- Very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Cholesterol (LDL)- Very high risk | -2.99 (26.243) | -23.41 (35.895) |  | -38.05 (38.867)
  Triglycerides- Low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Triglycerides- Low risk | -42.92 (48.340) | -28.67 (110.490) |  | -14.16 (35.044)
  Triglycerides- Moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Triglycerides- Moderate risk | 1.52 (43.420) | -22.32 (70.978) |  | -18.19 (61.094)
  Triglycerides- High risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Triglycerides- High risk | -3.85 (102.165) | -29.73 (116.182) | -83.19 (151.512) | -46.98 (127.625)
  Triglycerides- Very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Triglycerides- Very high risk | 23.34 (113.398) | -25.34 (102.889) |  | 4.47 (217.543)

6. Secondary Outcome: Percent Change From Baseline for Lipid Parameters at Week 12 Within Each CVD Risk Level
Description: Lipid parameters included LDL-C, High-Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol (TC), and Triglycerides (TG) according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes. The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Percent change from baseline was reported.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 1445 | 6 | 58
Percent Change
  Cholesterol- low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Cholesterol- low risk | -21.06 (18.145) | -15.39 (53.309) |  | -36.33 (23.292)
  Cholesterol- moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol- moderate risk | -11.66 (23.157) | -18.50 (24.651) |  | 73.60 (253.741)
  Cholesterol- high risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Cholesterol- high risk | -11.53 (24.302) | -13.91 (34.085) | -17.33 (19.989) | -15.34 (18.104)
  Cholesterol- very high risk: number analyzed (Participants) | 19 | 426 | 0 | 22
  Cholesterol- very high risk | 6.09 (22.562) | -11.07 (29.007) |  | -18.58 (24.524)
  Cholesterol (HDL) - low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Cholesterol (HDL) - low risk | 1.21 (15.236) | -1.55 (17.047) |  | -7.03 (35.153)
  Cholesterol (HDL)- moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol (HDL)- moderate risk | 4.08 (20.094) | 0.29 (18.265) |  | 12.12 (22.325)
  Cholesterol (HDL)- high risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Cholesterol (HDL)- high risk | 3.41 (29.176) | 4.59 (25.053) | 1.52 (15.985) | 2.42 (11.126)
  Cholesterol (HDL)- very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Cholesterol (HDL)- very high risk | 6.02 (22.796) | 6.55 (29.457) |  | -4.53 (13.600)
  Cholesterol (LDL)- low risk: number analyzed (Participants) | 12 | 127 | 0 | 2
  Cholesterol (LDL)- low risk | -31.33 (26.408) | -27.43 (22.633) |  | -47.37 (30.298)
  Cholesterol (LDL)- moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Cholesterol (LDL)- moderate risk | -18.59 (29.052) | -27.12 (27.917) |  | -20.86 (24.354)
  Cholesterol (LDL)- high risk: number analyzed (Participants) | 87 | 710 | 6 | 23
  Cholesterol (LDL)- high risk | -19.16 (32.501) | -21.81 (31.964) | -22.57 (26.524) | -20.59 (26.181)
  Cholesterol (LDL)- very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Cholesterol (LDL)- very high risk | 0.78 (34.076) | -12.68 (79.286) |  | -25.92 (25.288)
  Triglycerides- low risk: number analyzed (Participants) | 12 | 128 | 0 | 2
  Triglycerides- low risk | -21.40 (32.030) | -9.65 (39.610) |  | -9.63 (32.475)
  Triglycerides- moderate risk: number analyzed (Participants) | 21 | 145 | 0 | 9
  Triglycerides- moderate risk | 3.98 (40.156) | -8.81 (39.316) |  | -10.93 (37.268)
  Triglycerides- high risk: number analyzed (Participants) | 87 | 711 | 6 | 23
  Triglycerides- high risk | 13.35 (92.014) | -3.77 (50.582) | -27.55 (33.921) | -14.81 (34.606)
  Triglycerides- very high risk: number analyzed (Participants) | 19 | 425 | 0 | 22
  Triglycerides- very high risk | 36.01 (89.326) | -1.17 (62.412) |  | -10.55 (36.114)

7. Secondary Outcome: Study Drug Exposure for Overall - Total Dose and Week 12 Dose
Description: Atorvastatin total dose: calculated from Day 1 to Week 12 or last dose day; Week 12 dose: dose taken at Week 12
Time Frame: Day 1 to Week 12
Population: The analysis set included all participants who received at least 1 dose of atorvastatin. "Atorvastatin Unknown Dosage" did not have Week 12 dose. Number analyzed refers to number of participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
mg
  Total dose: number analyzed (Participants) | 291 | 3080 | 21 | 101 | 845
  Total dose | 958.90 (240.812) | 1816.63 (376.664) | 2506.19 (314.555) | 3326.93 (631.053) | 178.90 (136.33)
  Week 12 dose: number analyzed (Participants) | 280 | 2924 | 21 | 96 | 0
  Week 12 dose | 9.96 (0.422) | 20.00 (0.000) | 30.00 (0.000) | 40.00 (0.000) |

8. Secondary Outcome: Study Drug Exposure for Overall - Daily Dose
Description: Daily dose was calculated by total dose divided by the total days of receiving atorvastatin.
Time Frame: Day 1 to Week 12
Population: The analysis set included all participants who received at least 1 dose of atorvastatin and evaluable for specified category (daily dose).
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 845
mg/day | 10.43 (1.633) | 20.00 (0.423) | 29.00 (2.646) | 39.96 (0.314) | 20.09 (3.74)

9. Secondary Outcome: Study Drug Exposure Within Each CVD Risk Group - Total Dose and Week 12 Dose
Description: Atorvastatin total dose: calculated from Day 1 to Week 12 or last dose; Week 12 dose: dose taken at Week 12 according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Day 1 to Week 12
Population: The analysis set included all participants who received at least 1 dose of atorvastatin and only counted the participants at the dose levels: ≤10 mg, 20 mg, 30 mg and 40 mg. "Atorvastatin Unknown Dosage" arm within each CVD risk level was exclude since incomplete information on medication.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
mg
  Total dose (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Total dose (Low risk) | 975.00 (312.567) | 1760.84 (449.801) | 2790.00 (NA) — 1 participant of number analyzed | 3456.00 (1245.986)
  Total dose (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Total dose (Moderate risk) | 914.47 (224.965) | 1781.18 (415.197) | 2542.50 (261.964) | 3524.44 (464.519)
  Total dose (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Total dose (High risk) | 964.63 (254.036) | 1842.03 (383.312) | 2419.23 (342.332) | 3525.95 (373.954)
  Total dose (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Total dose (Very high risk) | 964.04 (152.396) | 1804.61 (328.691) | 2740.00 (96.437) | 3131.20 (685.669)
  Week 12 dose (Low risk): number analyzed (Participants) | 23 | 252 | 1 | 4
  Week 12 dose (Low risk) | 10.00 (0.000) | 20.00 (0.000) | 30.00 (NA) — 1 participant of number analyzed | 40.00 (0.000)
  Week 12 dose(Moderate risk): number analyzed (Participants) | 36 | 266 | 4 | 9
  Week 12 dose(Moderate risk) | 10.00 (0.000) | 20.00 (0.000) | 30.00 (0.000) | 40.00 (0.000)
  Week 12 dose (High risk): number analyzed (Participants) | 169 | 1419 | 13 | 37
  Week 12 dose (High risk) | 10.39 (1.678) | 20.00 (0.508) | 28.38 (3.254) | 39.97 (0.164)
  Week 12 dose (Very high risk): number analyzed (Participants) | 52 | 987 | 3 | 46
  Week 12 dose (Very high risk) | 10.00 (0.000) | 20.00 (0.000) | 30.00 (0.000) | 40.00 (0.000)

10. Secondary Outcome: Study Drug Exposure Within Each CVD Risk Group -Daily Dose
Description: Daily dose was calculated by total dose divided by the total days of receiving atorvastatin according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Day 1 to Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
mg/day
  Daily dose (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Daily dose (Low risk) | 10.81 (1.721) | 20.00 (0.000) | 30.00 (NA) — 1 participant of number analyzed | 40.00 (0.000)
  Daily dose (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Daily dose (Moderate risk) | 10.53 (1.572) | 20.03 (0.719) | 30.00 (0.000) | 40.00 (0.000)
  Daily dose (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Daily dose (High risk) | 10.39 (1.678) | 20.00 (0.508) | 28.38 (3.254) | 39.97 (0.164)
  Daily dose (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Daily dose (Very high risk) | 10.29 (1.486) | 20.00 (0.136) | 30.00 (0.000) | 39.94 (0.424)

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities and Treatment-related) for Overall
Description: All causalities adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage; Treatment-related AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; The event has a causal relationship with the treatment or usage.
Time Frame: Baseline to Week 12 (±28 days) or any unplanned visit (if occurred: any date during Week 4 to Week 16 )
Population: The Safety Analysis population included all participants who received at least 1 dose of study drug atorvastatin. Number analyzed refers to number of participants evaluable for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
Participants
  All causalities | 36 | 241 | 1 | 7 | 19
  Treatment-related | 17 | 107 | 1 | 2 | 6

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities and Treatment-related) by Dose Group Within Each CVD Risk Level
Description: All causalities adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage; Treatment-related AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; The event has a causal relationship with the treatment or usage. The AEs were categorized by the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline to Week 12 (±28 days) or any unplanned visit (if occurred: any date during Week 4 to Week 16 )
Population: The Safety Analysis population included all participants who received at least 1 dose of study drug atorvastatin and only counted the participants at the dose levels: ≤10 mg, 20 mg, 30 mg and 40 mg. "Atorvastatin Unknown Dosage" arm within each CVD risk level was exclude since incomplete information on medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
Participants
  All causalities (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  All causalities (Low risk) | 1 | 18 | 0 | 1
  All causalities (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  All causalities (Moderate risk) | 8 | 27 | 0 | 1
  All causalities (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  All causalities (High risk) | 22 | 126 | 1 | 1
  All causalities (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  All causalities (Very high risk) | 5 | 70 | 0 | 4
  Treatment-related (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Treatment-related (Low risk) | 0 | 7 | 0 | 0
  Treatment-related (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Treatment-related (Moderate risk) | 3 | 9 | 0 | 1
  Treatment-related (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Treatment-related (High risk) | 10 | 66 | 1 | 0
  Treatment-related (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Treatment-related (Very high risk) | 4 | 25 | 0 | 1

13. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) for Overall
Description: AESI were categorized as muscle symptoms: myalgia, fatigue, weakness, creatine kinase (CK) values 10 times the upper limit of normal, or rhabdomyolysis, and muscle damage based on significant elevated CK; major cardiovascular events: myocardial infarction, stroke, unstable angina requiring re-hospitalization, revascularization with either percutaneous coronary intervention or coronary-artery bypass grafting; Death.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred:any date during Week 4 to Week 16)
Population: The Safety Analysis population included all participants who received at least 1 dose of study drug atorvastatin.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
Participants | 18 | 146 | 1 | 5 | 7

14. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) by Dose Group Within Each CVD Risk Level
Description: AESI were categorized as muscle symptoms: myalgia, fatigue, weakness, creatine kinase (CK) values 10 times the upper limit of normal, or rhabdomyolysis, and muscle damage based on significant elevated CK; major cardiovascular events: myocardial infarction, stroke, unstable angina requiring re-hospitalization, revascularization with either percutaneous coronary intervention or coronary-artery bypass grafting; Death according to the CVD risk stratification. Low-risk: 10 years CV risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CV risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline (Day 1) to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
Participants
  Low risk: number analyzed (Participants) | 26 | 275 | 1 | 5
  Low risk | 1 | 9 | 0 | 0
  Moderate risk: number analyzed (Participants) | 38 | 287 | 4 | 9
  Moderate risk | 3 | 11 | 0 | 1
  High risk: number analyzed (Participants) | 175 | 1491 | 13 | 37
  High risk | 11 | 81 | 1 | 1
  Very high risk: number analyzed (Participants) | 52 | 1027 | 3 | 50
  Very high risk | 3 | 45 | 0 | 3

15. Secondary Outcome: Number of Participants With Elevated Abnormal Laboratory in Creatine Kinanse (CK), Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST) for Overall
Description: The elevated abnormal laboratory data was summarized: significant elevated CK: CK values 10 times the upper limit of normal; Persistent elevation in alanine aminotransferase, aspartate aminotransferase, or both: 2 consecutive measurements obtained 4 to 10 days apart that was more than 3 times the upper limit of the normal range.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
Participants
  ALT>3*ULN | 0 | 0 | 0 | 0 | 0
  AST>3*ULN | 0 | 0 | 0 | 0 | 0
  CK >= 10*ULN | 0 | 1 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Elevated Abnormal Laboratory in CK, ALT and AST by Dose Group Within Each CVD Risk
Description: The elevated abnormal laboratory data was summarized: significant elevated CK: CK values 10 times the upper limit of normal; Persistent elevation in alanine aminotransferase, aspartate aminotransferase, or both: 2 consecutive measurements obtained 4 to 10 days apart that was more than 3 times the upper limit of the normal range according to the CVD risk stratification. Low-risk: 10 years CV risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CV risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline to Week 12 (±28 days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
Participants
  ALT>3*ULN (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  ALT>3*ULN (Low risk) | 0 | 0 | 0 | 0
  ALT>3*ULN (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  ALT>3*ULN (Moderate risk) | 0 | 0 | 0 | 0
  ALT>3*ULN (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  ALT>3*ULN (High risk) | 0 | 0 | 0 | 0
  ALT>3*ULN (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  ALT>3*ULN (Very high risk) | 0 | 0 | 0 | 0
  AST>3*ULN (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  AST>3*ULN (Low risk) | 0 | 0 | 0 | 0
  AST>3*ULN (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  AST>3*ULN (Moderate risk) | 0 | 0 | 0 | 0
  AST>3*ULN (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  AST>3*ULN (High risk) | 0 | 0 | 0 | 0
  AST>3*ULN (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  AST>3*ULN (Very high risk) | 0 | 0 | 0 | 0
  CK >= 10*ULN (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  CK >= 10*ULN (Low risk) | 0 | 0 | 0 | 0
  CK >= 10*ULN (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  CK >= 10*ULN (Moderate risk) | 0 | 0 | 0 | 0
  CK >= 10*ULN (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  CK >= 10*ULN (High risk) | 0 | 1 | 0 | 0
  CK >= 10*ULN (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  CK >= 10*ULN (Very high risk) | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline for Clinical Laboratory Overall- ALT and AST
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from Baseline for ALT and AST date were reported.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
IU/L
  ALT-Week 12: number analyzed (Participants) | 141 | 1408 | 5 | 56 | 23
  ALT-Week 12 | 0.39 (25.362) | 1.60 (27.048) | 1.40 (8.414) | -0.25 (14.079) | -1.00 (21.058)
  ALT-Unplanned: number analyzed (Participants) | 34 | 239 | 1 | 4 | 9
  ALT-Unplanned | -0.04 (11.639) | 2.25 (17.861) | 5.00 (NA) — 1 participant of number analyzed | -20.70 (30.772) | 1.22 (13.000)
  AST- week 12: number analyzed (Participants) | 141 | 1396 | 5 | 56 | 22
  AST- week 12 | -1.50 (18.833) | -5.54 (47.298) | 3.60 (2.966) | -37.78 (87.382) | -17.48 (61.362)
  AST- unplanned: number analyzed (Participants) | 34 | 224 | 1 | 4 | 10
  AST- unplanned | -0.38 (6.605) | -8.43 (58.715) | 9.00 (NA) — 1 participant of number analyzed | -125.5 (184.247) | 2.22 (10.169)

18. Secondary Outcome: Change From Baseline for Clinical Laboratory Overall- Bilirubin, Blood Urea Nitrogen, Cholesterol, Creatinine, Triglycerides, Uric Acid
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from baseline for bilirubin, blood urea nitrogen, cholesterol (total), creatinine, triglycerides, uric acid data were reported.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
mg/dL
  Bilirubin-Week 12: number analyzed (Participants) | 136 | 1381 | 5 | 50 | 23
  Bilirubin-Week 12 | 0.02 (0.248) | 0.02 (0.323) | -0.01 (0.132) | 0.00 (0.301) | -0.08 (0.380)
  Bilirubin-Unplanned: number analyzed (Participants) | 34 | 236 | 1 | 3 | 9
  Bilirubin-Unplanned | -0.01 (0.301) | 0.04 (0.293) | 0.08 (NA) — 1 participant of number analyzed | -0.36 (0.190) | 0.09 (0.387)
  Blood urea nitrogen-Week 12: number analyzed (Participants) | 141 | 1366 | 5 | 57 | 21
  Blood urea nitrogen-Week 12 | 0.16 (5.238) | 0.10 (5.001) | -1.18 (2.989) | -0.29 (4.417) | -0.86 (9.287)
  Blood urea nitrogen- unplanned visit: number analyzed (Participants) | 35 | 216 | 1 | 4 | 10
  Blood urea nitrogen- unplanned visit | -1.18 (3.495) | -0.08 (5.326) | 3.11 (NA) — 1 participant of number analyzed | 4.66 (7.005) | -1.16 (3.911)
  Cholesterol- week 12: number analyzed (Participants) | 142 | 1417 | 6 | 56 | 20
  Cholesterol- week 12 | -26.13 (44.751) | -45.15 (393.221) | -40.35 (44.527) | -36.98 (54.175) | -27.20 (38.056)
  Cholesterol- unplanned visit: number analyzed (Participants) | 32 | 248 | 1 | 5 | 8
  Cholesterol- unplanned visit | -43.38 (31.472) | -55.38 (41.996) | -37.84 (NA) — 1 participant of number analyzed | -75.98 (56.967) | -24.23 (22.633)
  Creatinine- Week 12: number analyzed (Participants) | 142 | 1366 | 5 | 57 | 21
  Creatinine- Week 12 | 0.01 (0.202) | 0.01 (0.224) | -0.09 (0.158) | 0.00 (0.106) | 0.01 (0.165)
  Creatinine- unplanned: number analyzed (Participants) | 35 | 217 | 1 | 4 | 10
  Creatinine- unplanned | 0.00 (0.087) | 0.01 (0.130) | 0.01 (NA) — 1 participant of number analyzed | 0.09 (0.060) | -0.05 (0.131)
  Triglycerides- Week 12: number analyzed (Participants) | 142 | 1416 | 6 | 56 | 21
  Triglycerides- Week 12 | -3.95 (93.668) | -27.88 (108.151) | -83.19 (151.512) | -20.97 (160.296) | 8.22 (49.616)
  Triglycerides- unplanned: number analyzed (Participants) | 32 | 248 | 1 | 5 | 8
  Triglycerides- unplanned | -36.84 (67.068) | -46.19 (144.402) | -100.9 (NA) — 1 participant of number analyzed | -75.93 (88.578) | -25.67 (39.725)
  Uric acid- Week 12: number analyzed (Participants) | 140 | 1344 | 5 | 56 | 21
  Uric acid- Week 12 | -52.83 (621.039) | -0.08 (1.438) | -0.07 (0.795) | -0.20 (1.468) | -0.04 (1.781)
  Uric acid- unplanned visit: number analyzed (Participants) | 34 | 210 | 1 | 4 | 9
  Uric acid- unplanned visit | -0.29 (0.859) | 0.12 (1.159) | -0.30 (NA) — 1 participant of number analyzed | 0.68 (1.526) | -0.28 (0.957)

19. Secondary Outcome: Change From Baseline for Clinical Laboratory Overall- Creatine Kinase
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from Baseline for creatine kinase was reported.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
U/L
  Week 12: number analyzed (Participants) | 135 | 1264 | 5 | 54 | 16
  Week 12 | -12.77 (168.370) | -30.49 (388.838) | -7.60 (24.572) | -300.8 (698.733) | -139.0 (431.288)
  Unplanned visit: number analyzed (Participants) | 28 | 169 | 1 | 2 | 6
  Unplanned visit | 12.65 (59.880) | -26.74 (256.628) | 22.00 (NA) — 1 participant of number analyzed | -335.2 (469.795) | 23.67 (27.609)

20. Secondary Outcome: Change From Baseline for Clinical Laboratory by Dose Group Within Each CVD Risk Level-ALT and AST
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from Baseline for ALT and AST date were reported according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred:any date during Week 4 to Week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
IU/L
  ALT (Low risk)- Week 12: number analyzed (Participants) | 13 | 126 | 0 | 2
  ALT (Low risk)- Week 12 | -0.28 (14.557) | 1.68 (11.964) |  | 4.00 (15.556)
  ALT (Low risk)- unplanned visit: number analyzed (Participants) | 5 | 32 | 0 | 1
  ALT (Low risk)- unplanned visit | -2.80 (7.463) | 2.21 (15.514) |  | -29.23 (NA) — 1 participant of number analyzed
  ALT (moderate risk)- Week 12: number analyzed (Participants) | 22 | 142 | 0 | 9
  ALT (moderate risk)- Week 12 | -3.68 (15.438) | 0.83 (19.970) |  | 0.77 (6.612)
  ALT (moderate risk)- unplanned visit: number analyzed (Participants) | 5 | 21 | 0 | 0
  ALT (moderate risk)- unplanned visit | 0.00 (17.146) | -2.40 (16.196) |  |
  ALT (high risk)- Week 12: number analyzed (Participants) | 88 | 711 | 5 | 23
  ALT (high risk)- Week 12 | 5.27 (14.774) | 3.10 (31.018) | 1.40 (8.414) | 5.79 (11.825)
  ALT (high risk)- unplanned visit: number analyzed (Participants) | 20 | 106 | 1 | 0
  ALT (high risk)- unplanned visit | 0.99 (12.118) | 4.02 (12.412) | 5.00 (NA) — 1 participant of number analyzed |
  ALT(very high risk)- Week 12: number analyzed (Participants) | 18 | 429 | 0 | 22
  ALT(very high risk)- Week 12 | -17.98 (56.864) | -0.66 (25.035) |  | -7.36 (15.789)
  ALT(very high risk)- unplanned visit: number analyzed (Participants) | 4 | 80 | 0 | 3
  ALT(very high risk)- unplanned visit | -1.75 (8.382) | 1.14 (24.172) |  | -17.86 (37.039)
  AST (low risk)-Week 12: number analyzed (Participants) | 14 | 126 | 0 | 2
  AST (low risk)-Week 12 | -0.76 (9.684) | 0.76 (7.857) |  | 2.50 (7.778)
  AST (low risk)- unplanned visit: number analyzed (Participants) | 5 | 33 | 0 | 1
  AST (low risk)- unplanned visit | -1.00 (2.915) | -0.28 (6.874) |  | -8.56 (NA) — 1 participant of number analyzed
  AST (moderate risk)-Week 12: number analyzed (Participants) | 22 | 142 | 0 | 9
  AST (moderate risk)-Week 12 | -5.36 (16.276) | -1.49 (20.569) |  | -30.51 (92.532)
  AST (moderate risk)-unplanned visit: number analyzed (Participants) | 5 | 21 | 0 | 0
  AST (moderate risk)-unplanned visit | 2.80 (13.828) | -1.66 (5.743) |  |
  AST (high risk)-Week 12: number analyzed (Participants) | 88 | 708 | 5 | 23
  AST (high risk)-Week 12 | 1.89 (13.031) | -0.21 (21.587) | 3.60 (2.966) | 1.38 (7.432)
  AST (high risk)-unplanned visit: number analyzed (Participants) | 20 | 106 | 1 | 0
  AST (high risk)-unplanned visit | -0.75 (5.299) | 0.79 (12.214) | 9.00 (NA) — 1 participant of number analyzed |
  AST (very high risk)-Week 12: number analyzed (Participants) | 17 | 420 | 0 | 22
  AST (very high risk)-Week 12 | -14.62 (38.588) | -17.79 (79.278) |  | -85.34 (111.577)
  AST (very high risk)-unplanned visit: number analyzed (Participants) | 4 | 64 | 0 | 3
  AST (very high risk)-unplanned visit | -1.75 (3.862) | -30.13 (106.059) |  | -164.5 (204.461)

21. Secondary Outcome: Change From Baseline for Clinical Laboratory by Dose Group Within Each CVD Risk Level- Bilirubin, Blood Urea Nitrogen, Cholesterol, Creatinine, Triglycerides, Uric Acid
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from baseline for bilirubin, blood urea nitrogen, cholesterol (total), creatinine, triglycerides, uric acid data were reported according to the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
mg/dL
  Bilirubin (low risk)- Week 12: number analyzed (Participants) | 12 | 122 | 0 | 2
  Bilirubin (low risk)- Week 12 | -0.01 (0.237) | -0.03 (0.270) |  | 0.07 (0.167)
  Bilirubin (low risk)- unplanned visit: number analyzed (Participants) | 5 | 31 | 0 | 0
  Bilirubin (low risk)- unplanned visit | -0.07 (0.236) | 0.08 (0.225) |  |
  Bilirubin (moderate risk)- Week 12: number analyzed (Participants) | 22 | 139 | 0 | 9
  Bilirubin (moderate risk)- Week 12 | 0.02 (0.191) | 0.01 (0.305) |  | -0.09 (0.245)
  Bilirubin (moderate risk)- unplanned visit: number analyzed (Participants) | 5 | 21 | 0 | 0
  Bilirubin (moderate risk)- unplanned visit | -0.21 (0.237) | 0.01 (0.219) |  |
  Bilirubin (high risk)- Week 12: number analyzed (Participants) | 84 | 696 | 5 | 18
  Bilirubin (high risk)- Week 12 | 0.02 (0.271) | 0.03 (0.333) | -0.01 (0.132) | -0.04 (0.310)
  Bilirubin (high risk)- unplanned visit: number analyzed (Participants) | 20 | 105 | 1 | 0
  Bilirubin (high risk)- unplanned visit | 0.03 (0.294) | -0.01 (0.273) | 0.08 (NA) — 1 participant of number analyzed |
  Bilirubin (very high risk)- Week 12: number analyzed (Participants) | 18 | 424 | 0 | 21
  Bilirubin (very high risk)- Week 12 | 0.06 (0.209) | 0.02 (0.324) |  | 0.06 (0.324)
  Bilirubin (very high risk)- unplanned visit: number analyzed (Participants) | 4 | 79 | 0 | 3
  Bilirubin (very high risk)- unplanned visit | 0.07 (0.457) | 0.09 (0.350) |  | -0.36 (0.190)
  Blood urea nitrogen(low risk)-Week 12: number analyzed (Participants) | 14 | 121 | 0 | 2
  Blood urea nitrogen(low risk)-Week 12 | -1.08 (3.499) | 0.24 (2.990) |  | -2.38 (3.366)
  Blood urea nitrogen(low risk)-unplanned visit: number analyzed (Participants) | 4 | 26 | 0 | 1
  Blood urea nitrogen(low risk)-unplanned visit | -0.80 (0.783) | -0.98 (4.594) |  | -3.67 (NA) — 1 participant of number analyzed
  Blood urea nitrogen(moderate risk)-Week 12: number analyzed (Participants) | 21 | 137 | 0 | 9
  Blood urea nitrogen(moderate risk)-Week 12 | 1.18 (6.721) | -0.14 (3.887) |  | 1.56 (4.723)
  Blood urea nitrogen(moderate risk)-unplanned: number analyzed (Participants) | 5 | 18 | 0 | 0
  Blood urea nitrogen(moderate risk)-unplanned | -0.83 (2.386) | 1.91 (2.925) |  |
  Blood urea nitrogen(high risk)-Week 12: number analyzed (Participants) | 88 | 694 | 5 | 24
  Blood urea nitrogen(high risk)-Week 12 | 0.10 (5.191) | 0.20 (4.841) | -1.18 (2.989) | -0.99 (3.190)
  Blood urea nitrogen(high risk)-unplanned: number analyzed (Participants) | 22 | 98 | 1 | 0
  Blood urea nitrogen(high risk)-unplanned | -1.38 (4.248) | -0.36 (5.678) | 3.11 (NA) — 1 participant of number analyzed |
  cholesterol (low risk)-Week 12: number analyzed (Participants) | 13 | 133 | 0 | 2
  cholesterol (low risk)-Week 12 | -57.68 (46.926) | -47.63 (56.296) |  | -94.98 (71.530)
  cholesterol (low risk)-unplanned: number analyzed (Participants) | 5 | 34 | 0 | 1
  cholesterol (low risk)-unplanned | -47.41 (28.986) | -70.43 (46.727) |  | -122.8 (NA) — 1 participant of number analyzed
  cholesterol (moderate risk)-Week 12: number analyzed (Participants) | 22 | 145 | 0 | 9
  cholesterol (moderate risk)-Week 12 | -27.71 (41.919) | -43.23 (49.231) |  | -5.28 (61.380)
  cholesterol (moderate risk)-unplanned: number analyzed (Participants) | 4 | 21 | 0 | 0
  cholesterol (moderate risk)-unplanned | -44.59 (48.524) | -81.23 (42.498) |  |
  cholesterol (high risk)-week 12: number analyzed (Participants) | 88 | 713 | 6 | 23
  cholesterol (high risk)-week 12 | -27.72 (44.199) | -56.65 (551.937) | -40.35 (44.527) | -38.43 (49.029)
  cholesterol (high risk)-unplanned: number analyzed (Participants) | 19 | 114 | 1 | 0
  cholesterol (high risk)-unplanned | -42.78 (32.877) | -56.26 (39.587) | -37.84 (NA) — 1 participant of number analyzed |
  cholesterol (very high risk)-week 12: number analyzed (Participants) | 19 | 426 | 0 | 22
  cholesterol (very high risk)-week 12 | 4.63 (31.528) | -25.78 (49.060) |  | -43.16 (51.923)
  cholesterol (very high risk)-unplanned: number analyzed (Participants) | 4 | 79 | 0 | 4
  cholesterol (very high risk)-unplanned | -39.96 (15.081) | -40.75 (37.827) |  | -64.29 (58.435)
  creatinine (low risk)-Week 12: number analyzed (Participants) | 14 | 120 | 0 | 2
  creatinine (low risk)-Week 12 | 0.01 (0.119) | -0.01 (0.306) |  | 0.01 (0.007)
  creatinine (low risk)-unplanned: number analyzed (Participants) | 4 | 26 | 0 | 1
  creatinine (low risk)-unplanned | 0.01 (0.067) | 0.01 (0.146) |  | 0.14 (NA) — 1 participant of number analyzed
  creatinine (moderate risk)-Week 12: number analyzed (Participants) | 22 | 137 | 0 | 9
  creatinine (moderate risk)-Week 12 | -0.10 (0.299) | 0.00 (0.108) |  | -0.05 (0.081)
  creatinine (moderate risk)-unplanned: number analyzed (Participants) | 5 | 18 | 0 | 0
  creatinine (moderate risk)-unplanned | -0.07 (0.089) | -0.01 (0.101) |  |
  creatinine (high risk)-Week 12: number analyzed (Participants) | 88 | 694 | 5 | 24
  creatinine (high risk)-Week 12 | 0.02 (0.175) | 0.01 (0.201) | -0.09 (0.158) | 0.00 (0.120)
  creatinine (high risk)- unplanned: number analyzed (Participants) | 22 | 98 | 1 | 0
  creatinine (high risk)- unplanned | 0.00 (0.091) | -0.01 (0.137) | 0.01 (NA) — 1 participant of number analyzed |
  creatinine (very high risk)- Week 12: number analyzed (Participants) | 18 | 415 | 0 | 22
  creatinine (very high risk)- Week 12 | 0.09 (0.200) | 0.01 (0.258) |  | 0.02 (0.102)
  creatinine (very high risk)-unplanned: number analyzed (Participants) | 4 | 75 | 0 | 3
  creatinine (very high risk)-unplanned | 0.04 (0.053) | 0.03 (0.119) |  | 0.08 (0.062)
  triglycerides (low risk)- week 12: number analyzed (Participants) | 13 | 133 | 0 | 2
  triglycerides (low risk)- week 12 | -45.48 (47.189) | -31.41 (114.297) |  | -14.16 (35.044)
  triglycerides (low risk)- unplanned: number analyzed (Participants) | 5 | 34 | 0 | 1
  triglycerides (low risk)- unplanned | 21.42 (28.999) | -75.82 (101.162) |  | -188.5 (NA) — 1 participant of number analyzed
  triglycerides (moderate risk)- week 12: number analyzed (Participants) | 22 | 145 | 0 | 9
  triglycerides (moderate risk)- week 12 | 0.00 (42.967) | -22.32 (70.978) |  | -18.19 (61.094)
  triglycerides (moderate risk)- unplanned: number analyzed (Participants) | 4 | 21 | 0 | 0
  triglycerides (moderate risk)- unplanned | -32.08 (14.674) | -53.27 (61.766) |  |
  triglycerides (high risk)- week 12: number analyzed (Participants) | 88 | 713 | 6 | 23
  triglycerides (high risk)- week 12 | -4.70 (101.889) | -29.87 (116.122) | -83.19 (151.512) | -46.98 (127.625)
  triglycerides (high risk)- unplanned: number analyzed (Participants) | 19 | 114 | 1 | 0
  triglycerides (high risk)- unplanned | -47.56 (70.510) | -54.85 (189.895) | -100.9 (NA) — 1 participant of number analyzed |
  triglycerides (very high risk)- week 12: number analyzed (Participants) | 19 | 425 | 0 | 22
  triglycerides (very high risk)- week 12 | 23.34 (113.398) | -25.34 (102.889) |  | 4.47 (217.543)
  triglycerides (very high risk)- unplanned: number analyzed (Participants) | 4 | 79 | 0 | 4
  triglycerides (very high risk)- unplanned | -63.50 (89.174) | -19.08 (85.039) |  | -47.79 (71.981)
  uric acid (low risk)-Week 12: number analyzed (Participants) | 14 | 120 | 0 | 2
  uric acid (low risk)-Week 12 | -0.33 (0.838) | -0.06 (0.980) |  | 0.32 (0.933)
  uric acid (low risk)-unplanned: number analyzed (Participants) | 4 | 26 | 0 | 1
  uric acid (low risk)-unplanned | -0.13 (0.337) | 0.23 (1.139) |  | 0.00 (NA) — 1 participant of number analyzed
  uric acid (moderate risk)-Week12: number analyzed (Participants) | 20 | 138 | 0 | 9
  uric acid (moderate risk)-Week12 | -0.84 (2.753) | -0.16 (1.335) |  | -0.61 (1.285)
  uric acid (moderate risk)-unplanned: number analyzed (Participants) | 5 | 18 | 0 | 0
  uric acid (moderate risk)-unplanned | -0.87 (0.833) | -0.47 (1.493) |  |
  uric acid (high risk)-week 12: number analyzed (Participants) | 88 | 683 | 5 | 23
  uric acid (high risk)-week 12 | -0.38 (1.875) | -0.07 (1.447) | -0.07 (0.795) | -0.58 (1.664)
  uric acid (high risk)-unplanned: number analyzed (Participants) | 21 | 96 | 1 | 0
  uric acid (high risk)-unplanned | -0.13 (0.879) | -0.16 (1.047) | -0.30 (NA) — 1 participant of number analyzed |
  uric acid (very high risk)-week 12: number analyzed (Participants) | 18 | 403 | 0 | 22
  uric acid (very high risk)-week 12 | -407.9 (1732.170) | -0.05 (1.568) |  | 0.32 (1.237)
  uric acid (very high risk)-unplanned: number analyzed (Participants) | 4 | 70 | 0 | 3
  uric acid (very high risk)-unplanned | -0.55 (1.039) | 0.60 (1.051) |  | 0.90 (1.786)
  Blood urea nitrogen (Very high risk)- Week 12: number analyzed (Participants) | 18 | 414 | 0 | 22
  Blood urea nitrogen (Very high risk)- Week 12 | 0.21 (4.794) | -0.03 (5.975) |  | -0.09 (5.417)
  Blood urea nitrogen (Very high risk)- unplanned: number analyzed (Participants) | 4 | 74 | 0 | 3
  Blood urea nitrogen (Very high risk)- unplanned | -0.89 (1.766) | 0.12 (5.484) |  | 7.43 (5.237)

22. Secondary Outcome: Change From Baseline for Clinical Laboratory by Dose Group Within Each CVD Risk Level- Creatine Kinase
Description: The baseline data was collected within 1 month before taking atorvastatin or within 24 hours after starting atorvastatin. Change from Baseline for creatine kinase was reported according to the CVD risk stratification. Low-risk: 10 years CV risk <5%; Moderate-risk: 10 years CVD risk 5%~10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CV risk 10%~15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
U/L
  Creatine Kinase(Low risk-Week 12: number analyzed (Participants) | 11 | 116 | 0 | 2
  Creatine Kinase(Low risk-Week 12 | 15.40 (47.148) | 22.89 (135.208) |  | 15.75 (22.274)
  Creatine Kinase(Low risk-unplanned visit: number analyzed (Participants) | 4 | 25 | 0 | 0
  Creatine Kinase(Low risk-unplanned visit | 3.00 (16.793) | 29.41 (112.521) |  |
  Creatine Kinase(moderate risk)-Week 12: number analyzed (Participants) | 22 | 126 | 0 | 8
  Creatine Kinase(moderate risk)-Week 12 | 0.45 (46.688) | 0.03 (73.412) |  | -363.4 (1078.110)
  Creatine Kinase(moderate risk)-unplanned visit: number analyzed (Participants) | 1 | 14 | 0 | 0
  Creatine Kinase(moderate risk)-unplanned visit | 8.00 (NA) — 1 participant of number analyzed | 6.76 (30.302) |  |
  Creatine Kinase(high risk)-Week 12: number analyzed (Participants) | 85 | 641 | 5 | 22
  Creatine Kinase(high risk)-Week 12 | -1.99 (118.333) | 14.49 (209.095) | -7.60 (24.572) | -0.25 (18.669)
  Creatine Kinase(high risk)-unplanned visit: number analyzed (Participants) | 19 | 88 | 1 | 0
  Creatine Kinase(high risk)-unplanned visit | 10.96 (62.211) | 3.17 (87.977) | 22.00 (NA) — 1 participant of number analyzed |
  Creatine Kinase(very high risk)-Week 12: number analyzed (Participants) | 17 | 381 | 0 | 22
  Creatine Kinase(very high risk)-Week 12 | -102.0 (387.028) | -132.5 (637.616) |  | -607.2 (800.209)
  Creatine Kinase(very high risk)-unplanned visit: number analyzed (Participants) | 4 | 42 | 0 | 2
  Creatine Kinase(very high risk)-unplanned visit | 31.50 (90.246) | -134.0 (479.298) |  | -335.2 (469.795)

23. Secondary Outcome: Precentage of Participants With Discontinuation From the Study for Overall
Description: Percentage of participants who dropped out of the study and reasons for discontinuation were summarized overall.
Time Frame: 12 weeks of follow-up
Population: as for outcome 11
Measure: Number; unit: Percent
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
Number analyzed (Participants) | 291 | 3080 | 21 | 101 | 1055
Percent
  Death | 0 | 0.03 | 0 | 0 | 0.37
  Relation to study drug not defined | 0.68 | 1.10 | 0 | 2.97 | 96.77
  AE Related to study drug | 0 | 0.03 | 0 | 0 | 0.47
  AE Not related to study drug | 0.34 | 0 | 0 | 0 | 0.37

24. Secondary Outcome: Precentage of Participants With Discontinuation From the Study by Dose Group Within Each CVD Risk Level
Description: Percentage of participants who dropped out of the study and reasons for discontinuation were summarized by the CVD risk stratification. Low-risk: 10 years CVD risk <5%; Moderate-risk: 10 years CVD risk 5% to 10%; High-risk: Coronary Heart Disease (CHD) or CHD risk equivalents, or 10 years CVD risk 10% to 15%; Very-high risk: acute coronary syndromes, or ischemic cardiovascular disease combined with diabetes.
Time Frame: 12 weeks of follow-up
Population: as for outcome 12
Measure: Number; unit: Percent
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 291 | 3080 | 21 | 101
Percent
  Death (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Death (Low risk) | 0 | 0 | 0 | 0
  Relation to study drug not defined (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Relation to study drug not defined (Low risk) | 0 | 0.36 | 0 | 20.0
  Related to study drug (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Related to study drug (Low risk) | 0 | 0.36 | 0 | 0.32
  Not related to study drug (Low risk): number analyzed (Participants) | 26 | 275 | 1 | 5
  Not related to study drug (Low risk) | 0 | 0 | 0 | 0
  Death (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Death (Moderate risk) | 0 | 0 | 0 | 0
  Relation to study drug not defined (Moderate risk): number analyzed (Participants) | 291 | 287 | 4 | 9
  Relation to study drug not defined (Moderate risk) | 0 | 2.43 | 0 | 0
  Related to study drug (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Related to study drug (Moderate risk) | 0 | 0 | 0 | 0
  Not related to study drug (Moderate risk): number analyzed (Participants) | 38 | 287 | 4 | 9
  Not related to study drug (Moderate risk) | 0 | 0 | 0 | 0
  Death (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Death (High risk) | 0 | 0.06 | 0 | 0
  Relation to study drug not defined (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Relation to study drug not defined (High risk) | 1.14 | 1.07 | 0 | 2.70
  Related to study drug (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Related to study drug (High risk) | 0 | 0 | 0 | 0
  Not related to study drug (High risk): number analyzed (Participants) | 175 | 1491 | 13 | 37
  Not related to study drug (High risk) | 0.57 | 0 | 0 | 0
  Death (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Death (Very high risk) | 0 | 0 | 0 | 0
  Relation to study drug not defined(Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Relation to study drug not defined(Very high risk) | 0 | 0.97 | 0 | 2.00
  Related to study drug (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Related to study drug (Very high risk) | 0 | 0 | 0 | 0
  Not related to study drug (Very high risk): number analyzed (Participants) | 52 | 1027 | 3 | 50
  Not related to study drug (Very high risk) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 12 (±28 Days) or any unplanned visit (if occurred: any date during Week 4 to Week 16)
Arm/Group | Atorvastatin <=10 mg | Atorvastatin 20 mg | Atorvastatin 30 mg | Atorvastatin 40 mg | Atorvastatin Unknown Dosage
All-Cause Mortality (participants affected / at risk) | 0/291 | 2/3080 | 0/21 | 0/101 | 5/1055
Serious Adverse Events (participants affected / at risk) | 5/291 | 68/3080 | 0/21 | 3/101 | 9/1055
Other Adverse Events (participants affected / at risk) | 0/291 | 0/3080 | 0/21 | 0/101 | 0/1055
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin <=10 mg (N=291) | Atorvastatin 20 mg (N=3080) | Atorvastatin 30 mg (N=21) | Atorvastatin 40 mg (N=101) | Atorvastatin Unknown Dosage (N=1055)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pelvic mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitations of the study are intrinsic to its observational, non-controlled, non-randomized design. This study stopped enrollment prior to meeting the planned sample size and was not committed to submit to China agency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT02565615/SAP_000.pdf
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT02565615/Prot_001.pdf